CLINICAL TRIAL: NCT05059808
Title: European Sepsis Care Survey
Status: Completed | Type: Observational
Sponsor: University Medicine Greifswald (Other)
Collaborators: European Sepsis Alliance (Unknown); European Society of Anaesthesiology and Intensive Care (Other); European Society for Emergency Medicine (EUSEM) Research Network (Network); European Society of Clinical Microbiology and Infectious Diseases, ESGBIES Study Group (Unknown); European Society of Intensive Care Medicine (Other); Sepsisdialog, Germany (Unknown); European Shock Society (Unknown); Becton, Dickinson and Company (Industry)
Responsible Party: Principal Investigator, Christian S. Scheer, MD, Principle Investigator, University Medicine Greifswald
Other Study IDs: ESA_Survey01; BB 124/21 (Other: Ethics Committee University Medicine Greifswald)
Record Dates: First submitted 2021-08-31; First posted 2021-09-28 (Actual); Last update posted 2023-06-13 (Actual); Status verified 2023-06

CONDITIONS: Sepsis
MeSH Terms: conditions — Sepsis

STUDY DESIGN:
Observational Model: Other | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
The objective of this survey is to investigate the current state of sepsis care around Europe. The study is aiming at hospital structure, emergency departments, wards, intensive care units and clinical diagnostic and microbiological service.

ELIGIBILITY:
Inclusion Criteria:

* Hospitals of all strata

Exclusion Criteria:

-

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: European hospitals
Sampling Method: Non-Probability Sample
Enrollment: 1450 (Actual)
Dates: Start 2021-08-01 (Actual); Primary Completion 2022-04-30 (Actual); Study Completion 2022-10-30 (Actual)

PRIMARY OUTCOMES:
Questionnaire | 2021
  Structure of sepsis care in Europe

CONTACTS AND LOCATIONS:
Overall Officials: Christian S Scheer, Principal Investigator — Anesthesiology and Intensive Care Medicine Department, University of Greifswald, Germany; Adam Linder, Principal Investigator — European Sepsis Alliance; Daniela Filipescu, Principal Investigator — European Sepsis Alliance, European Society of Anaesthesiology and Intensive Care; Evangelos Giamarellos-Bourboulis, Principal Investigator — European Sepsis Alliance, European Shock Society; Evgeny Idelevich, Principal Investigator — ESCMID/Study Group for Bloodstream Infections, Endocarditis and Sepsis; Konrad Reinhart, Principal Investigator — Global Sepsis Alliance; Matthias Gründling, Principal Investigator — Quality management project Sepsisdialog; Ricard Ferrer, Principal Investigator — European Society of Intensive Care Medicine; Said Laribi, Principal Investigator — European Society for Emergency Medicine (EUSEM) Research Network; Manu Malbrain, Principal Investigator — International Fluid Academy; Gabriella Bottari, Principal Investigator — European Society of Paediatric and Neonatal Intensive Care
Locations (20):
- Emergency Department Antwerp University Hospital, Edegem, Belgium
- Department of Anesthesiology and Intensive Care Medicine University Hospital of Ostrava, Ostrava-Poruba, Czechia
- Department of Emergency Medicine University of Southern Denmark, Odense, Denmark
- Perioperative, Intensive Care and Pain Medicine Helsinki University Hospital, Helsinki, Finland
- Hopital Raymond Poncare Service de Reanimation Medicale, Garches, France
- University Medicine Greifswald, Greifswald, Germany
- 4th Department of Internal Medicine ATTIKON University Hospital, Athens, Greece
- National Institute for Antibiotic Resistance & Infection Control, Ministry of Health, Tel Aviv, Israel
- Ospedale Niguarda Ca' Granda Milano, Milan, Italy
- State University of Medicine and Pharmaceutics "Nicolae Testemiţanu", Chisinau, Moldova
- University Medical Center Groningen, Groningen, Netherlands
- St Olavs hospital, Trondheim, Norway
- Department of Anaesthesiology and Intensive Therapy Wroclaw Medical University, Wroclaw, Poland
- Universidade do Porto Faculdade de Medicina: Porto, Porto, Portugal
- "Prof CC Iliescu" Emergency Institute for Cardiovascular Diseases, Bucharest, Bucharest, Romania
- Vladimir L. Vanevskii Department of Anaesthesiology and Reanimatology, North-Western State Medical University named after Ilya I. Mechnikov, Saint Petersburg, Russia
- Corporació Sanitària Parc Taulí · critical care center, sabadell hospital, Corporació Sanitaria Universitaria Parc Tauli, Sabadell, Spain
- Faculty of Medicine, Department of Clinical Sciences Lund, Division of Infection Medicine, Lund University, Lund, Sweden
- Hacettepe University, Department of Internal Medicine Sihhiye, Ankara, Ankara, Turkey (Türkiye)
- King's College London, Guy's and St Thomas' Foundation Hospital, Department of Critical Care, London, London, United Kingdom

IPD SHARING:
Plan to Share IPD: No
This study uses no patient data.

REFERENCES:
- [Derived] Ceccato A, Scheer CS, Ferrer R, Martinez ML, Cistero B, Yebenes JC, Trenado J, Lorencio C, Linder A, Filipescu D, Idelevich EA, Giamarellos-Bourboulis EJ, Artigas A; European Sepsis Care Study Group. Regional sepsis care in Catalonia: comparative insights from a secondary analysis of the European Sepsis Care Survey. Crit Care. 2025 Aug 19;29(1):367. doi: 10.1186/s13054-025-05507-3. No abstract available. PMID 40830495